CLINICAL TRIAL: NCT02290275
Title: Creatine, Exercise and Inflammatory Markers in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Dr. Stephen Mark Cornish, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2014:117
Record Dates: First submitted 2014-11-10; First posted 2014-11-14 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Creatine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): The subjects in this arm will receive 20 grams of a placebo (maltodextrin) for 1 week and then 5 grams of placebo (maltodextrin) for 11 weeks in addition to their regular diets.
  Interventions: Dietary Supplement: placebo (maltodextrin)
- Creatine (Experimental): The subjects in this arm will receive 20 grams of creatine for 1 week and then 5 grams of creatine for 11 weeks in addition to their regular diets.
  Interventions: Dietary Supplement: Creatine
- Walking Exercise (Experimental): The subjects in this arm will receive a walking exercise program on a motorized treadmill where they will walk for 30 minutes at 3.1 mph, 3 days per week for 12 weeks.
  Interventions: Other: Walking Exercise

INTERVENTIONS:
Dietary Supplement: Creatine — Subjects will supplement their regular diet with 20 grams of creatine for 1 week and then 5 grams of creatine for the following 11 weeks.
  Arms: Creatine
Other: Walking Exercise — Subjects will walk on a specialized treadmill that lowers the impact of walking by taking up to 80% of their body weight away. The subjects will exercise by walking on this treadmill at 3.1 mph, 3 days per week for 30 minutes per day for 12 weeks.
  Arms: Walking Exercise
Dietary Supplement: placebo (maltodextrin) — Subjects will supplement their regular diet with 20 grams of maltodextrin for 1 week and then 5 grams of maltodextrin for the following 11 weeks.
  Arms: Placebo

SUMMARY:
The goal of this research project is to determine the effectiveness of creatine supplementation and supported low-load walking exercise for managing systemic inflammatory biomarkers and joint symptoms in individuals diagnosed with chronic symptomatic knee osteoarthritis. The central hypothesis of this investigation is that creatine supplementation and exercise will significantly lower systemic biomarkers of inflammation in patients diagnosed with knee osteoarthritis.

DETAILED DESCRIPTION:
Participants will provide informed consent, complete participant information and knee demographic forms, and undergo radiographic evaluation to confirm eligibility. Baseline evaluation of (1) systemic inflammation; and (2) knee joint pain and function will be completed. Following baseline evaluation, participants will be randomly assigned to 1 of 3 groups using online software available at http://www.randomizer.org/:

1. Exercise group: Participants will exercise for 30 minutes under low-load walking conditions 3x per week for 12 consecutive weeks on a Lower Body Positive Pressure (LBPP) treadmill (Alter-G Inc - Menlo Park, CA) at a set speed of 3.1 mph at 0⁰ incline. The initial five minutes of each exercise session will be used as a warm-up to allow the participant to reach their target heart rate, to accommodate to walking on the treadmill's belt surface, and to facilitate adjustment of the LBPP within the treadmill's air chamber to a percentage of unweighting that eliminates or substantially reduces the participant's acute knee pain for the duration of the 30 minute walking session. Subjects will be blinded to the amount of LBPP used to un-weight them during each low-load walking session.
2. Creatine group: Participants will supplement their regular diet with creatine monohydrate for 12 consecutive weeks. In week #1, participants will ingest 5 grams of creatine monohydrate 4x per day for a total ingestion of 20 grams per day. For the remaining 11 weeks, participants will consume 5 grams of creatine monohydrate per day to maintain the increased concentration of creatine.
3. Placebo group: Participants in the placebo group will supplement their regular diet with maltodextrin (an inert sugar based molecule) for 12 consecutive weeks. In week #1, participants will ingest 5 grams of maltodextrin 4x per day for a total ingestion of 20 grams per day. They will then ingest 5 grams of maltodextrin per day for the remaining 11 weeks.

All data collection will take place at the Pan Am Clinic, a multidisciplinary tertiary care hospital and research facility that serves as the Winnipeg Regional Health Authority's "Centre of Excellence for Musculoskeletal Injury Assessment and Treatment". This project will utilize the combined assets of University of Manitoba and Pan Am Clinic to access medical resources that are used on a daily basis for the diagnosis, treatment, and long term management of patients with knee OA. All participants will undergo follow-up evaluation 13 weeks after their initial baseline evaluation.

Aim #1: Determine if knee OA systemic inflammation is significantly decreased following completion of a 12 week creatine supplementation or low-load treadmill walking exercise regimen.

Hypotheses:

* There will be a significant decrease in systemic inflammation following completion of a 12 week creatine supplementation program.
* There will be a significant decrease in systemic inflammation following completion of a 12 week low-load walking exercise program.
* There will be no decrease in systemic inflammation following completion of a 12 week placebo supplementation program.

Primary Outcome Measures: Systemic inflammation will be evaluated by obtaining venous blood samples from the participants. Blood samples (approximately 20 mL) will be drawn by venipuncture from the antecubital vein into cooled (4°C) vacutainer tubes containing EDTA under sterile conditions. After inversion, tubes will be centrifuged at 1065g for 15 minutes at 4°C. Approximately 8 mL of plasma will be aliquoted into Eppendorf tubes (8 x 1 mL per tube) and frozen at -80°C until analysis. All plasma samples will be evaluated for C-reactive protein, interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α), interleukin-1β (IL-1β), and interleukin-10 (IL-10) using an enzyme linked immunosorbent assay (ELISA) kit according to the manufacturer's instructions. All assays will be analyzed in duplicate within the same microplate to reduce variation. Serum will be obtained by drawing a blood sample by venipuncture into vacutainer serum separator tubes. This serum will be used to analyze the serum cartilage oligomeric matrix protein (sCOMP) using an ELISA kit according to the manufacturer's instructions.

Aim #2: Determine if knee OA joint pain and function are significantly altered following completion of a 12 week creatine supplementation or low-load treadmill walking exercise regimen.

Hypotheses:

* There will be a significant decrease in knee OA joint pain and dysfunction following completion of a 12 week creatine supplementation program.
* There will be a significant decrease in knee OA joint pain and dysfunction following completion of a 12 week low-load walking exercise program.
* There will be no significant decrease in knee OA joint pain and dysfunction following completion of a 12 week placebo supplementation program.

Primary Outcome Measures: Knee pain during normal activities of daily living (ADLs) will be evaluated using the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire. The KOOS is a self-administered, knee-specific questionnaire that is designed to measure OA patient's knee pain over the previous seven-day period. Testing indicates that it is a valid, highly reliable and responsive measurement tool for evaluating changes after different OA interventions.

Secondary Outcome Measures: Bilateral knee joint function and physical health will be evaluated through the following measures both pre and post study:

1. Goniometric assessment of knee joint range of motion (ROM) is a clinically accepted procedure for evaluating joint function. It allows the reliable and accurate quantification of movement using linear (cm) and angular units (degrees).
2. Isokinetic evaluation of thigh muscle strength is the gold standard method used to quantify thigh muscle strength about an OA knee joint in both longitudinal and clinical investigations, as well as to examine the effect of creatine or exercise interventions on patients with knee OA.
3. Measurement of cardiovascular (CV) capacity via maximum volume of oxygen uptake (VO2 max) testing. VO2 max testing assesses the maximum amount of oxygen that a person can consume per minute at a maximum work rate and is considered the best measure of cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* (1) Ages 45-65; (2) Body mass index (BMI) over 25 kg/m2; (3) Knee pain when performing normal activities of daily living (walking, squatting, or kneeling); (4) Kellgren & Lawrence grades II & III radiographic evidence of mild to moderate knee osteoarthritis in one or both knees.

Exclusion Criteria:

* (1) Radiographic evidence of severe knee osteoarthritis; (2) History of traumatic hip, knee, or ankle injury or surgery; (3) Use of crutches or a walking aid during ambulation; (3) History of medical conditions that prevent physical activity; (4) Unable to provide consent due to language barrier or mental status; (5) History of diabetes, cardiovascular disease, or screen positive for ankylosing spondylitis, psoriatic arthritis, chronic reactive arthritis, or renal problems requiring peritoneal dialysis or hemodialysis; (6) Unwillingness or inability to return for follow-up appointments.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
C-reactive protein | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cornish, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Alison Longo, Winnipeg, Manitoba, Canada